CLINICAL TRIAL: NCT03347266
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injection for Post-operative Pain Following Total Hip Arthroplasty
Brief Title: Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injection for Postoperative Pain Following Total Hip Arthroplasty.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT-VVZ149-06
Record Dates: First submitted 2017-11-06; First posted 2017-11-20 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2017-11

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VVZ-149 injections (Experimental): VVZ-149 injections will be mixed with saline, then intravenous infusion for 10hr. The drug product will be administrated with a 1000mg for 10 hours.
  Interventions: Drug: VVZ-149 injections
- Placebo (Placebo Comparator): Placebo group will receive an water for injection the same volume and period of experimental group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149 injections — •VVZ-149 injection
  Other Names: Colorless, transparent liquid in water for injection
  Arms: VVZ-149 injections
Drug: Placebo — water for injection
  Other Names: water for injection
  Arms: Placebo

SUMMARY:
The purpose of this phase 2 study is to evaluate the efficacy and safety of an analgesic drug candidate, VVZ-149 Injections. The study is designed as randomized, double-blind, parallel, and placebo-controlled study.

DETAILED DESCRIPTION:
VVZ-149 is a dual antagonist of GlyT2 and 5HT2A. GlyT2 blockage increases inhibitory synaptic transmission by glycine in the spinal cord, resulting in a reduction of pain transmissions to the brain. 5HT2A blockage decreases descending serotonergic facilitatory modulation on pain transmission by the brain and reduces nociceptor activation in peripheral nerves, which are primary sources of pain in post-surgical pain. VVZ-149 has been shown to have comparable efficacy to morphine in well controlled (blind, complete randomization with a positive control) animal studies using rat models of post-operative pain and formalin-induced pain. The PK/PD study in animals indicates that therapeutic plasma concentration in human subjects will be 600-1,900 ng/ml. A clinical Phase 1 study performed in healthy subjects has shown no clinically significant adverse events up to a plasma concentration level of 3,261 ng/ml other than brief symptoms of mild nausea or dizziness, and mild somnolence when the plasma exposure level is more than 2,000 ng/ml.

ELIGIBILITY:
Inclusion Criteria:

1. Patient between the ages of 25 and 65 years old
2. Male patient, in the case of female patient, postmenopausal women, or women physically incapable of childbearing
3. Subject who underwent surgery specially for the clinical study
4. Ability to provide written informed consent prior to any study procedures.
5. Ability to understand study procedures and communicate clearly with the investigator and staff.
6. Subjects with body weight under 100kg and body mass index (BMI) level lower than 35 kg/m2, inclusive
7. Single-side surgery patient

Exclusion Criteria:

< Surgical Factors >

1. Emergency or unplanned surgery.
2. Repeat operation

   < Subject Characteristics >
3. Women with childbearing potential, Women who are pregnant or breastfeeding.
4. Unstable or poorly controlled psychiatric condition (e.g., untreated PTSD, anxiety, or depression). Subjects who take stable doses of antidepressants and anti-anxiety drugs may be included.
5. Unstable or acute medical condition (e.g., unstable angina, congestive heart failure, renal failure, hepatic failure, AIDS).
6. Subjects who have long QPR (>200msec) or prolonged QTc (> 450msec in male, >470msec in female) at Screening

   < Drug, Alcohol, and Pharmacological Considerations >
7. History of alcohol, opiate or other drug abuse or dependence within 12 months prior to Screening .
8. Ongoing or recent (within 6 hour prior to surgery) use of steroids, opioids, or antipsychotics.
9. Alcohol consumption within 24 hours of surgery.
10. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) or acetaminophen within 6 hours of surgery.
11. Use of herbal agents or nutraceuticals (i.e., chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian) within 7 days prior to surgery.

    < Anesthetic and Other Exclusion Considerations >
12. Use of neuraxial or regional anesthesia related to the surgery.
13. Use of ketamine, gabapentin, pregabalin, or lidocaine (>1 mg/kg) intra or peri-operatively, or within 24 hours of surgery.
14. Subject with known allergies to hydromorphone.
15. Subjects who received another investigational drug within 30 days of scheduled surgery

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Change of Pain Intensity | prior to PCA, at 0,1, 2, 4, 6, 8, 10, 24 hours post-PCA
  Change of Pain Intensity assessed using the Numerical Rating Scale (NRS, 0-10)

SECONDARY OUTCOMES:
Fentanyl Consumption | 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-16, 16-18, 18-20, 20-22, 22-24 hours post-PCA
  the amount of fentanyl consumption over 24 hours
the number of Fentanyl request | 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-16, 16-18, 18-20, 20-22, 22-24 hours post-PCA
  the number of PCA request over 24 hours
the amount of rescue dose | 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-16, 16-18, 18-20, 20-22, 22-24 hours post-dose
  the amount of rescue dose over 24 hours
the number of requested rescue dose | 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-16, 16-18, 18-20, 20-22, 22-24 hours post-dose
  the amount of requested rescue dose over 24 hours
Area under a curve (AUC) of Pain intensity and sum of AUC of pain intensity (SPI) | 0-1, 1-2, 2-4, 4-6, 6-8, 8-10, 10-24 hours post-PCA
  the calculated AUC of Pain intensity and sum of AUC of pain intensity (SPI)
Global measurement of patient satisfaction assessed on the questionnaire (0-5 points scale) | 8, 24 hours post-PCA
  the assessment of global satisfaction of patients using 0-5 points scale
the correlation between Pharmacokinetic (PK) and Pharmacodynamic (PD) | 0, 2, 6 hours post-PCA
  Correlation between total opioid consumption (fentanyl dose equivalents) and plasma exposure of study drug at 0, 2, 6 hours post-PCA
Number of Vomiting | 8, 24 hours post-PCA
  the number of vomiting after PCA

CONTACTS AND LOCATIONS:
Overall Officials: Seonjun Bae, MD, PhD, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea